CLINICAL TRIAL: NCT04549324
Title: Sleep Apnea, Coronary Atherosclerosis and Heart Failure in Diabetes Patients With Nephropathy
Acronym: SLEEP
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-122-20
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2021-10

CONDITIONS: Sleep Apnea; Diabetic Nephropathy Type 2; Coronary Atheroscleroses; Heart Insufficiency; Arterial Stiffness; Kidney Diseases; Vascular Diseases
MeSH Terms: conditions — Sleep Apnea Syndromes; Coronary Artery Disease; Heart Failure; Kidney Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood, Plasma, Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sleep Apnea (AHI ≥ 15 per hour): Patients with moderate/severe sleep apnea (Apnea/hypopnea-index ≥ 15 per hour).
- Non-Sleep Apnea (AHI < 5 per hour): Patients without sleep apnea (Apnea/hypopnea-index < 5 per hour).

SUMMARY:
Background:

Diabetes, and especially diabetic kidney disease is associated with the development of cardiovascular disease such as calcification in the coronary arteries and heart failure. Sleep apnea is frequent among patients with diabetes and diabetic kidney disease and sleep apnea itself is a solitary risk factor in the development of cardiovascular disease. Nonetheless, sleep apnea is underdiagnosed in diabetes patients because of a discrepancy between sleep apnea severity and actual oxygen deficiency symptoms which makes the diagnosis difficult. For that reason, many diabetics have undiagnosed sleep apnea together with cardiovascular disease. Early discovery of sleep apnea among high risk diabetic patients may therefore be considered crucial before cardiovascular complications develop. For this reason, sleep apnea screening of high-risk diabetics can possibly improve early diagnostics of cardiovascular disease.

Aim:

This study will seek to establish the association between obstructive sleep apnea (OSA) and coronary calcification and heart failure in patients with diabetic kidney disease. The basic hypothesis of the study is that patients with diabetic kidney disease and concurrent OSA have a higher prevalence and severity of coronary calcification and heart failure compared to patients without OSA.

Methods:

Diabetic adult patients with scheduled check-ups at Steno Diabetes Center Aarhus, or Department of Renal Medicine on Aarhus University Hospital will be included in the study.

Firstly, all included patients are screened for sleep apnea with the devices SomnoTouch® and ApneaLink®. Based on the sleep apnea determination; 40 patients with moderate-severe sleep apnea are compared with 40 patients without sleep apnea. In both groups, the patients are examined for calcification in the coronary vessels using a CT-scan while the function of the heart is examined by ultrasound (echocardiography). The stiffness of aorta is measured and performed using radial artery tonometry (SphygmoCor®).

Furthermore, range of blood- and urine samples will be performed

The perspectives are that patients with diabetes should be regularly evaluated for sleep apnea and that patients with moderate/severe sleep apnea should undergo further examination for cardiovascular disease even though the patients don't display any symptoms of either cardiovascular disease or sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years.
* Diabetes Mellitus Type 2 with an eGFR between 10-60 ml/min/1,73 m^2 (Equalling CKD-group 3, 4 and 5 non-dialysis).

Exclusion Criteria:

* Known sleep apnea in continuous positive airway pressure(CPAP) treatment.
* Known mild sleep apnea (AHI 5-14) after the sleep apnea measurement.
* Participants with central apnea (> 50 % of central apnea episodes in the AHI ≥ 15 group.) or Cheyne Stokes after the sleep apnea measurement.
* < 4 hours of recording (ApneaLink)
* Known coronary arterial disease with previous revascularization (PCI or CABG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic adult patients (Type 2) with scheduled check-ups at Steno Diabetes Center Aarhus, or Department of Renal Medicine on Aarhus University Hospital can be included in the study if they satisfy all eligible criteria. Additionally, patients from the GP and within the including area of Aarhus University Hospital were invited to participate in the study.
  The study cohort will consist of:
  Generel characteristics of both groups:
  - Diabetes Mellitus Type 2 with an eGFR between 10-60 ml/min/1,73 m^2
  Sleep Apnea:
  1. 40 patients with an apnea/hyponea-index above ≥ 15 per hour.
     Non-Sleep Apnea:
  2. 40 patients with an apnea/hyponea-index below < 5 per hour.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
The association between sleep apnea and coronary atherosclerosis (Agatston Score) measured with cardiac CT-scan in patients with diabetic nephropathy. | Cardiac CT-scan will be performed no later than 1 month after inclusion. All Agatston scores will be estimated straight after the cardiac CT-scan.
  The degree of atherosclerosis in the coronary artery walls is evaluated by cardiac CT-scan and subsequent quantified by Agatston score. Patients with an estimated glomerular filtration rate (eGFR) ≤ 25 ml/min/1,73 m2 is scanned without contrast whereas patients with an eGFR 26-60 ml/min/1,73 m2 are screened with contrast.
  All Agatston scoring will be performed by a cardiologist blinded to information on patient biochemical characteristics and AHI. The only biochemical parameter which the cardiologist is not blinded to is eGFR.
The association between sleep apnea and systolic function in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in the study will undergo transthoracic echocardiography. Systolic function is evaluated by two-dimensional automated evaluation of ejection fraction (2-D auto-EF).
  The echocardiographic-clinician is blinded to AHI-status.
The association between sleep apnea and diastolic heart failure in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in the study will undergo transthoracic echocardiography. Diastolic function is evaluated by E/e´.
  The echocardiographic-clinician is blinded to AHI-status.
The association between sleep apnea and systolic function in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in the study will undergo transthoracic echocardiography. Systolic function is evaluated by Left Ventricular Global Longitudinal Strain (GLS).
  The echocardiographic-clinician is blinded to AHI-status.

SECONDARY OUTCOMES:
The association between sleep apnea and coronary plaque volume in patients with diabetic nephropathy. | Cardiac CT-scan will be performed no later than 1 month after inclusion.
  Coronary plaque volume is estimated by a cardiac CT-scan with contrast.
  All coronary plaque volume analysing will be performed by a cardiologist blinded to information on patient biochemical characteristics and AHI. The only biochemical parameter which the cardiologist is not blinded to is eGFR.
Association of sleep apnea and aortic stiffness (defined as Pulse Wave Velocity (PWV)) in patients with diabetic nephropathy. | PWV is performed the same day as the patient is included.
  To get a non-invasive estimate of the aortic stiffness, measurement of Pulse Wave Velocity (PWV) (carotid-femoral and carotid-radial) will be performed. PWV will be recorded with the Sphygmocor® device according to regular protocol. If possible, two acceptable measurements will be conducted for each included patient. Calculation of PWV will be performed automatically by the device using a previously published formula.
Association between Matrix Gla Protein (MGP) and coronary calcification in patients with sleep apnea and diabetic nephropathy. | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in patients with sleep apnea and diabetic nephropathy. MGP, a novel biochemical marker of arterial calcification, will be collected and analysed in all patients.
Association between Calcification propensity score (T50test) and coronary calcification in patients with sleep apnea and diabetic nephropathy. | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in patients with sleep apnea and diabetic nephropathy. Calcification propensity score (T50test) will be collected and analysed in all patients.
Association between sRANKL (soluble receptor activator of nuclear factor kappa-B ligand) and coronary calcification in patients with sleep apnea and diabetic nephropathy. | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in patients with sleep apnea and diabetic nephropathy. sRANKL (soluble receptor activator of nuclear factor kappa-B ligand) will be collected and analysed in all patients.
Association between 25-OH-Vitamin D(D3+D2) and coronary calcification in patients with sleep apnea and diabetic nephropathy. | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in patients with sleep apnea and diabetic nephropathy. 25-OH-Vitamin D(D3+D2) will be collected and analysed in all patients.
Association between Fetuin-A(alfa-2-Heremans Schmid glycoprotein; AHSG) and coronary calcification in patients with sleep apnea and diabetic nephropathy. | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021.
  To establish a deeper understanding of the pathogenesis of central arterial calcification in patients with sleep apnea and diabetic nephropathy. Fetuin-A(alfa-2-Heremans Schmid glycoprotein; AHSG) will be collected and analysed in all patients
Association between Sclerostin and coronary calcification in patients with sleep apnea and diabetic nephropathy. | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in patients with sleep apnea and diabetic nephropathy., Sclerostin will be collected and analysed in all patients
Association between osteoprotegerin and coronary calcification in patients with sleep apnea and diabetic nephropathy. | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in patients with sleep apnea and diabetic nephropathy., osteoprotegerin will be collected and analysed in all patients.
Association between BsAP (bone-specific alkaline phosphatase) and coronary calcification in patients with sleep apnea and diabetic nephropathy. | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in patients with sleep apnea and diabetic nephropathy., BsAP (bone-specific alkaline phosphatase) will be collected and analysed in all patients
Association between TRAP5B (tartrate-resistant acid phosphatase 5b) and coronary calcification in patients with sleep apnea and diabetic nephropathy. | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in patients with sleep apnea and diabetic nephropathy, TRAP5B (tartrate-resistant acid phosphatase 5b) will be collected and analysed in all patients.
Association between P1NP (procollagen type 1 N propeptide) and coronary calcification in patients with sleep apnea and diabetic nephropathy. | Analysis will be performed as batch-analysis at the end of inclusion of patients summer 2021
  To establish a deeper understanding of the pathogenesis of central arterial calcification in patients with sleep apnea and diabetic nephropathy., P1NP (procollagen type 1 N propeptide) will be collected and analysed in all patients
Association between LVEDd (Left ventricular end diastolic diameter) as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between LVEDs (Left ventricular end systolic diameter) as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between IVSd (Interventricular Septal Thickness at Diastole) as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between IVSs (Interventricular Septal Thickness at Systole) as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between PWTd (Posterior wall thickness at end-diastole) as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between PWTs (Posterior wall thickness at end-systole) as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between Aorta (sinus valsalva) diameter as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between Aorta (Ascendens) diameter as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between Aorta (Abdominalis) diameter as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between maximum Vena Cava Inferior diameter as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between minimum Vena Cava Inferior diameter as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between Early mitral inflow velocity (E) as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between Late mitral inflow velocity (A) as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between E/A-ratio as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between Deceleration time of early diastolic transmittal flow (dtE) as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between Right ventricular diameter (RVD) as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus.
  The echocardiographic-clinician is blinded to AHI-status.
Association between left atrial volume (LAV) as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. The echocardiographic-clinician is blinded to AHI-status.
Association between 2D atrial global strain as determined during echocardiography and sleep apnea in patients with diabetic nephropathy. | Transthoracic echocardiography will be performed no later than 1 month after inclusion and prior to cardiac CT-scan
  All patients included in this study will undergo echocardiography. In particular systolic and diastolic function will be in focus. The echocardiographic-clinician is blinded to AHI-status.

CONTACTS AND LOCATIONS:
Overall Officials: Niels H. Buus, MD PhD DMSc, Study Chair — Department of Renal diseases, Aarhus University Hospital; Sebastian Nielsen, MD student, Principal Investigator — Department of Renal diseases, Aarhus University Hospital; Jakob T. Nyvad, MD, Study Chair — The Clinic of Hypertension, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD. pas